CLINICAL TRIAL: NCT00000678
Title: Dideoxycytidine ( Ro 24-2027 ) A Randomized, Open-Label, Comparative Study of Dideoxycytidine ( ddC ) Versus Zidovudine ( AZT ) in Patients With AIDS or Advanced ARC Who Have Received Long-Term AZT Therapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Hoffmann-La Roche (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 119; N3492B
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 1992-09

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Drug Evaluation; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine; Zalcitabine

INTERVENTIONS:
Drug: Zidovudine
Drug: Zalcitabine

SUMMARY:
To compare the effectiveness of zalcitabine ( dideoxycytidine; ddC ) therapy to zidovudine ( AZT ) in the treatment of AIDS or advanced AIDS related complex ( ARC ) in patients who have already received at least 1 year of AZT therapy and to define the safety profile.

ddC has been shown to have an antiviral effect, and AZT is known to significantly decrease mortality and to reduce the frequency of opportunistic infections in patients with AIDS or advanced ARC. After 1 year of AZT therapy, the effectiveness tends to diminish and patients progress with more opportunistic infections and higher mortality rates. This may be due to the emergence of AZT resistant virus isolated from some patients who have been on long-term AZT therapy. These isolates were still sensitive to ddC. A study of long-term effectiveness of ddC in patients with AIDS or advanced ARC who have been on long-term AZT therapy is warranted because (1) ddC has antiviral activity, (2) there is no blood toxicity associated with taking ddC, and (3) the effectiveness of ddC in test tube studies does not seem to be diminished by decreased effectiveness of AZT.

DETAILED DESCRIPTION:
ddC has been shown to have an antiviral effect, and AZT is known to significantly decrease mortality and to reduce the frequency of opportunistic infections in patients with AIDS or advanced ARC. After 1 year of AZT therapy, the effectiveness tends to diminish and patients progress with more opportunistic infections and higher mortality rates. This may be due to the emergence of AZT resistant virus isolated from some patients who have been on long-term AZT therapy. These isolates were still sensitive to ddC. A study of long-term effectiveness of ddC in patients with AIDS or advanced ARC who have been on long-term AZT therapy is warranted because (1) ddC has antiviral activity, (2) there is no blood toxicity associated with taking ddC, and (3) the effectiveness of ddC in test tube studies does not seem to be diminished by decreased effectiveness of AZT.

AMENDED: AZT will be administered orally every 4 or 5 hours. Patients in the second arm discontinue AZT and take ddC as two tablets every 8 hours. Duration of the study is 1 year with interim analysis done at 6 months after 75 percent enrollment and at end of the study. Original design: Patients with AIDS or advanced ARC who have been receiving at least 500 mg/day of AZT for at least 48 weeks are randomized to 1 of 2 treatment arms. Patients in the first treatment arm continue their current dose of AZT.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Aerosolized pentamidine will be given, as tolerated for all patients, for Pneumocystis carinii pneumonia prophylaxis at a dose of 300 mg once every 4 weeks.

Allowed maintenance treatment with:

* Pyrimethamine (= or < 75 mg/day).
* Sulfadiazine (< 4 gl/day).
* Amphotericin (1 mg/kg/day up to 5 days).
* Fluconazole (400 mg/day).
* Ketoconazole (400 mg/day).
* Acyclovir (up to 12.4 mg/kg q8h IV for zoster or up to 4000 mg/day will be allowed PO with precautions - nausea and vomiting possible with doses > 1000 mg/day).
* Ganciclovir (6 mg/kg/day).
* Medications for tuberculosis or Mycobacterium avium for patients who have recovered from toxoplasmosis, cryptococcosis, candidiasis, herpes virus infections, cytomegalovirus infections, tuberculosis, or Mycobacterium avium intracellulare.
* Erythropoietin and megace as needed.
* Isoniazid if patient has no peripheral neuropathy at study entry and is taking pyridoxine at least 50 mg/day concomitantly.
* Phenytoin if patient has no peripheral neuropathy at study entry and has been stable on the drug for at least 3 months.

Patients must have had Pneumocystis carinii pneumonia (PCP) and no other AIDS defining opportunistic infection present when zidovudine (AZT) therapy was first initiated.

Patients must have:

* Advanced AIDS related complex (ARC).
* Antibody to HIV by federally licensed ELISA and confirmed by Western blot analysis.
* Ability to give conformed consent.

Exclusion Criteria

Co-existing Condition:

Patients are excluded who:

* Have had zidovudine (AZT) therapy interrupted for > 30 consecutive days at any time during AZT therapy or have been off AZT for > 90 days total.
* Have had AZT therapy interrupted for "recurrent" grade 4 toxicity, defined as > one episode of the same grade 4 toxicity after dose interruption or attenuation.
* Have visceral or extensive Kaposi's sarcoma requiring therapy or any other malignancy requiring therapy.
* Have a history of peripheral neuropathy.

Concurrent Medication:

Excluded:

* Other experimental medications, including foscarnet, ribavirin, and fluconazole (prior to IND approval).
* Other antiretroviral agents, biologic modifiers or corticosteroids.
* Drugs that can cause peripheral neuropathy including phenytoin (under conditions not specifically allowed), hydralazine, metronidazole, nitrofurantoin, vincristine, cisplatinum, dapsone, disulfiram, and diethyldithiocarbamate.

Patients with the following are excluded:

* History of peripheral neuropathy or moderate to severe peripheral neuropathy as defined by the combination of signs or symptoms of peripheral neuropathy and findings indicative of peripheral neuropathy on the standardized neurologic exam.
* Active opportunistic infection.
* Participation in another research treatment study.

Prior Medication:

Excluded:

* Dideoxycytidine (ddC).
* Didanosine (ddI).

Active substance or alcohol abuse.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320
Dates: Primary Completion 1992-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Davies Med Ctr, San Francisco, California
  - Mount Zion Med Ctr, San Francisco, California
  - Univ of Miami School of Medicine, Miami, Florida
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Albany Med College / AIDS Treatment Ctr, Albany, New York
  - Holmes Hosp / Univ of Cincinnati Med Ctr, Cincinnati, Ohio
  - Graduate Hosp, Philadelphia, Pennsylvania
  - N Texas Ctr for AIDS & Clin Rsch, Dallas, Texas

REFERENCES:
- [Background] Fischl MA, Olson RM, Follansbee SE, Lalezari JP, Henry DH, Frame PT, Remick SC, Salgo MP, Lin AH, Nauss-Karol C, Lieberman J, Soo W. Zalcitabine compared with zidovudine in patients with advanced HIV-1 infection who received previous zidovudine therapy. Ann Intern Med. 1993 May 15;118(10):762-9. doi: 10.7326/0003-4819-118-10-199305150-00002. PMID 8097082
- [Background] Gries JM, Troconiz IF, Verotta D, Jacobson M, Sheiner LB. A pooled analysis of CD4 response to zidovudine and zalcitabine treatment in patients with AIDS and AIDS-related complex. Clin Pharmacol Ther. 1997 Jan;61(1):70-82. doi: 10.1016/S0009-9236(97)90183-1. PMID 9024175